CLINICAL TRIAL: NCT00658151
Title: Ultrasound Diagnosis of Antibiotic Associated Diarrhea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Radiologist, Shaare Zedek Medical Center
Other Study IDs: avital.ctil
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Antibiotic-Associated Diarrhea
Keywords: focus; study; evaluate; sonographic; findings; colon; patients; developed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The hypothesis is that there are unique sonographic characteristics of antibiotic-associated diarrhea. We will compare the ultrasound findings in patients who received antibiotics and developed diarrhea to toxin analysis for clostridium difficile in stool in order to find differences in the sonographic findings in the positive and negative cases.

ELIGIBILITY:
Inclusion Criteria:

* admitted patients who developed diarrhea in 72 hours since the beginning of admission
* patients age above 18 years.
* patients received antibiotics during admission

Exclusion Criteria:

* other reasons of diarrhea
* drugs induced diarrhea
* length of time since the beginning of diarrhea is shorter than 72 hours.
* patients had diarrhea during the first day of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in internal and geriatrics departments who developed diarrhea in a period of 72 hours since the beginning of admission and received antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel